CLINICAL TRIAL: NCT04246593
Title: Effectiveness and Implementation of a Research Tested Mobile Produce Market Designed to Improve Diet in Underserved Communities
Brief Title: Effectiveness and Implementation of a Research Tested Mobile Produce Market
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lucia A Leone, Assistant Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1144594; 5R37CA215232-02 (NIH)
Record Dates: First submitted 2019-10-22; First posted 2020-01-29 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Fruit and Vegetable Consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Market (Experimental): Partner sites that are randomized to the "Intervention - Market" will plan and start (or expand) a Mobile Market and run the Market weekly for at least 10 months (non necessarily nonconsecutive). The Mobile Market will follow the Veggie Van Model which includes a "share model", price reductions (incentives), and an educational component.
  Interventions: Other: Mobile Market program implementation
- Control - Planning (No Intervention): At Control - Planning (comparison) sites, engagement will focus on involving community members in food access program planning and research. It is anticipated that each organization will create one or more community advisory committees to oversee their food access work. At comparison sites, engagement efforts will be more generally centered on food access and understanding what types of programs would be most acceptable. Examples of community engagement activities include community forums and listening sessions, informational tables at community events, and establishment of text, e-mail or social media sites for ongoing communication and feedback around food access issues. As part of this community engagement work, partners will collect contact information from community members that will assist in the data collection process.

INTERVENTIONS:
Other: Mobile Market program implementation — Mobile Market program implementation includes utilizing a Veggie Van model which sells reduced cost locally-grown produce in communities with barriers to accessing fresh F&Vs because of availability, cost, or lack of produce preparation skills.The Veggie Van visits sites that already serve the target market (e.g., lower-income housing communities, community health centers, community colleges). While Mobile Market programs vary in their model and operation, we believe that the three components of Veggie Van's success are it's "share" model, price reductions (incentives), and educational component
  Arms: Intervention - Market

SUMMARY:
Investigators will test the effectiveness of the Veggie Van model across multiple organizations and sites using a cluster-randomized design and will document the implementation process to understand what factors are associated with dietary change and sustainability.

DETAILED DESCRIPTION:
After 9 qualified organizations have been identified among applicants, investigators will randomize proposed Mobile Market (MM) sites (33 total across all partner organizations), to an intervention (Mobile Market program implementation) or comparison condition (extended planning). Randomization will be stratified within each organization so that each organization will have 2 intervention and 2 comparison sites. One organization will have 5 sites. The 5th site will allow for more thorough testing of protocol procedures. This ensures that study groups will be balanced at the organizational level. The condition for which each proposed MM location was selected will be communicated at the time of award. Organizations will communicate to intervention sites that they want to open a MM at that location within the next year. Organizations will communicate to comparison sites that they want to work with them on a food systems planning process to determine if a MM program is the right fit for their location. At the end of the year-long planning process with comparison sites, the organization and proposed MM site will decide together how to proceed (start a MM, apply for grant funding for a different project; etc.).

Both arms will undergo community engagement efforts that serve to both identify potential research participants and engage them in the planning for a MM. Intervention sites will work with a community advisory committee to develop an engagement plan to raise community awareness of the forthcoming MM.

Comparison sites will work with a community advisory committee to engage community members in a food access planning process.

Both intervention and comparison sites will distribute interest forms as part of the community engagement process.Research staff will identify from the interest forms those interested in participating in the study. Consent will be obtained via phone. Phone surveys and in-person data collection will then be completed.

* Baseline and 12 month Follow-Up Survey will include dietary-related psychosocial measures These surveys will be administered over the phone.
* The main individual-level outcome, change in Fruits and Veggies (F&V) intake at 12 months, will be measured through four 24-hour recalls (2 at baseline and 2 at 12 months) which will be administered over the phone by trained interviewers. One recall at each time point will be from a weekday and the other from a weekend day. Recalls will be collected using the Nutrition Data Systems for Research (NDSR) computer-based software application. A participant will receive The Food Amounts Booklet via mail after the baseline survey to have as a visual reference for the 24-hour recalls.
* In addition to survey data, body mass index (BMI) and dermal carotenoids will be measured at in-person data collection events at baseline and 12 months.

Market (Intervention Sites) will implement a Mobile Market, weekly, for at least 10 months that will follow the Veggie Van model that includes 3 research supported components:

* "Share" model: Similar to community supported agriculture, this model selects fresh, high quality produce available from local farmers, creates "shares" of 5-8 types of produce, and delivers to community sites once per week. Customers can also choose to purchase individual produce items; however, based on focus group discussions with customers, it is believed that the share model is a key factor in increasing consumption of a larger quantity and variety of Fruits and Veggies. It also contributes to program sustainability by allowing Mobile Markets to better predict their sales and reduce waste.
* Incentives: Prices for a Veggie Van model vary slightly by market location. In some communities, only one reduced price (i.e., lower than market value) is offered. In other communities, where customers are of mixed socioeconomic status, partners offer shares on a sliding scale. Customers can use their ebt card, credit/debit, cash or check to purchase produce shares. To support the subsidized cost of produce for low-income residents, the Veggie Van model offers a full-cost box delivery service to workplaces and schools. However, other communities may be able to take advantage of incentive programs (such as Double Up Food Bucks) to offer reduced costs to those eligible.
* Educational Component: The Veggie Van model has a curriculum that consists of monthly themes (e.g., Eating in Season, Healthy Snacks, MyPlate, Reducing Sugar) and weekly lessons which build upon those themes. The lessons are designed to be delivered at the Mobile Market while customers are on line waiting to make a purchase. Accompanying newsletters help reinforce lesson plans and also include information about storing and preparing the produce items in the box that week. Newsletters include seasonal recipes and when possible, cooking demonstrations of these recipes or taste tests of featured produce items are offered at the Mobile Market Partner site.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old, speak English or Spanish
* the primary grocery shopper for their household
* interested in having more healthy food retail options at or around the proposed Mobile Market site
* either frequent the proposed Mobile Market site regularly or live near by

Exclusion Criteria:

* Individuals will be excluded if they do not meet the above inclusion criteria. They will be excluded if they are planning to leave the area or stop using the proposed Mobile Market site (intervention participants) within the next year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Leone, Phd, Principal Investigator — SUNY at Buffalo
Locations (1):
- Massachusetts Avenue Project, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leone LA, Kasprzak C, Lally A, Paluch R, Haynes-Maslow L, Raja S, Tumiel-Berhalter L, Vermont LN, Ammerman A. Cluster-Randomized Controlled Trial of a Mobile Produce Market designed to Address Diet and Food Insecurity in Underserved Communities. Res Sq [Preprint]. 2025 Dec 2:rs.3.rs-7860050. doi: 10.21203/rs.3.rs-7860050/v1. PMID 41377950
- [Derived] Vermont LN, Kasprzak C, Lally A, Claudio A, Tumiel-Berhalter L, Haynes-Maslow L, Ammerman A, Raja S, Leone LA. A Randomized Controlled Trial of a Research-Tested Mobile Produce Market Model Designed to Improve Diet in Under-Resourced Communities: Rationale and Design for the Veggie Van Study. Int J Environ Res Public Health. 2022 Aug 10;19(16):9832. doi: 10.3390/ijerph19169832. PMID 36011468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-based organizations selected as study partners facilitated participant recruitment through a 2-month community engagement period prior to the intervention. If recruitment goals were not met, recruitment continued for up to two months after the intervention period started. Intervention/delayed-intervention control activities occurred at partner sites on a rolling basis; the first participant was enrolled January 13, 2020 and the last was enrolled September 25, 2022.
Pre-assignment Details: Of 759 eligible participants enrolled in the study, 699 were included in analysis as 60 participants were removed because the partner organization operating the intervention/delayed-intervention control sites they were assigned to dropped out of the study.
Period: Overall Study
Arm/Group | Intervention - Market | Control - Planning
Started | 426 | 273
Completed | 281 | 186
Not Completed | 145 | 87
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Lost to Follow-up | 124 | 71
Not completed — Moved out of area/became ineligible | 3 | 1
Not completed — Reason unknown | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Market | Control - Planning | Total
Number analyzed (Participants) | 426 | 273 | 699
Age, Categorical [Count of Participants; unit: Participants] — Population: Number of participants analyzed is different from the overall population due to missing data from survey responses.
  Participants
    number analyzed (Participants) | 409 | 256 | 665
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 359 | 197 | 556
    >=65 years | 50 | 59 | 109
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 64 | 43 | 107
  Female | 359 | 230 | 589
  Other/Refused/Missing | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 21 | 73
  Not Hispanic or Latino | 374 | 252 | 626
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 174 | 150 | 324
  White | 189 | 92 | 281
  More than one race | 17 | 10 | 27
  Unknown or Not Reported | 30 | 15 | 45
Region of Enrollment [Number; unit: participants]
  United States | 426 | 273 | 699
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.58 (7.46) | 31.91 (8.34) | 31.1 (7.83)

OUTCOME MEASURES:

1. Primary Outcome: Consumption of Fruits and Vegetables
Description: Change in Fruit & Vegetable (F&V) intake (servings/day) at 12 months will be calculated from four 24-hour recalls (2 at baseline and 2 at 12-months) which will be administered over the phone by trained interviewers (in English or Spanish). One recall at each time point will be from a weekday and the other from a weekend day. The 24-hour dietary recalls will be collected using the Nutrition Data Systems for Research (NDSR) computer-based software application developed at the University of Minnesota Nutrition Coordinating Center (NCC); NDSR uses a five pass interview approach with interview prompts in English and Spanish (49). The NCC Food and Nutrient Database serves as the source of food composition information in NDSR (50). When a participant completes their in-person data collection, participants will receive The Food Amounts Booklet to have as a visual reference during the 24-hour recall. This booklet is compatible with the NDSR program.
Time Frame: 12 months
Population: The food environment and shopping behaviors were significantly impacted by the COVID-19 pandemic in 2020. Many intervention participants did not attend the mobile market. We analyzed the data according to participants' self-reported intervention usage. We combined intervention participants who reported never using the intervention with the Control - Planning (comparison) arm participants, as these participants all did not receive/use the intervention.
Measure: Mean (Standard Error); unit: servings/day
Groups:
- Mobile Market Intervention Users: Many study participants that were randomized to the Intervention - Market arm of this study reported not attending the mobile market at least once; this is largely attributable to the significant impact of the COVID-19 pandemic in 2020, the year this study began recruitment. 171 intervention participants self-reported shopping at the Veggie Van at least once (40.1%).
- Mobile Market Intervention Non-Users: Non-users include both those participants who were randomized to the intervention arm that reported never attending the Veggie Van mobile market intervention combined with those participants who were randomized to the Control - Planning (comparison) arm. These participants never received the intervention.
Arm/Group | Mobile Market Intervention Users | Mobile Market Intervention Non-Users
Number analyzed (Participants) | 171 | 369
servings/day | -0.24 (0.44) | -0.13 (0.28)
Statistical Analysis 1: Comparison: Mobile Market Intervention Users vs Mobile Market Intervention Non-Users; Test type: Other — We used generalized linear mixed model (GLMM) with random intercept to control for clustering within sites. In order to further explore the intervention effect, we fit GLMMs that adjust for (1) baseline dietary intake and (2) race and baseline income; p = 0.84, GLMM — P-value calculated for the mean difference between the user and non-user groups; Mean Difference (Final Values) = -0.11, Standard Error of Mean 0.52

2. Secondary Outcome: Body Mass Index
Description: BMI will be calculated at baseline and 12 months from weight measured using a Seca 876 digital scale (maximum capacity of 250 kg) and height measured to the nearest 1/8 inch using a Seca stadiometer. Weight and height will be combined to report BMI in kg/m^2
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Change in mean kg/m^2
Arm/Group | Intervention - Market | Control - Planning
Number analyzed (Participants) | 42 | 34
Change in mean kg/m^2 | -0.05 (0.77) | -0.54 (0.86)
Statistical Analysis 1: Comparison: Intervention - Market vs Control - Planning; Test type: Other — We used generalized linear mixed model (GLMM) with random intercept to control for clustering within sites; p = 0.61, GLMM — P-value calculated for the mean difference between change in BMI for intervention and control groups; Median Difference (Net) = -0.59, Standard Error of Mean 1.15

3. Secondary Outcome: Dermal Carotenoids
Description: Dermal Carotenoids will be measured using a finger scan technology called the "Veggie Meter" which relies on pressure mediated Raman Spectroscopy (RS) and is thought to be a valid indicator of changes in skin carotenoids in response to dietary carotenoid consumption. Dermal Carotenoids are measured on a scale of 0 to 800, with 0 representing the absence of dermal carotenoids and 800 representing the maximum possible score for dietary carotenoids. A higher dermal carotenoid score indicates a greater presence of dietary carotenoids, and as such a better outcome. Change between baseline and follow-up scores will be calculated for each group.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Market | Control - Planning
Number analyzed (Participants) | 42 | 33
score on a scale | -22.19 (29.89) | 5.83 (31.35)
Statistical Analysis 1: Comparison: Intervention - Market vs Control - Planning; Test type: Other — We used generalized linear mixed model (GLMM) with random intercept to control for clustering within sites; p = 0.53, GLMM — P-value calculated for the mean difference in change scores between the intervention and control groups; Mean Difference (Net) = -28.02, Standard Error of Mean 43.31

4. Other Pre Specified Outcome: Psychosocial Measures - Self-efficacy
Description: Self-efficacy to purchase, prepare and eat fresh F&V were measured using a 10-point Likert scale, where 10 indicates easiest (most self-efficacy, better outcome) and 1 indicates hardest (least self-efficacy, worse outcome), applied to a selection of 8 items adapted from a study of shoppers where self-efficacy was shown to be correlated with nutrition behaviors and will serve as a comprehensive assessment of the effect of the educational intervention. The 8 items' scores were summed to create a total self-efficacy score ranging from 8 (least total self-efficacy, worse outcome) to 80 (most total self-efficacy, better outcome) for each participant. The measured outcome is the difference between the mean baseline total self-efficacy score and the mean follow-up total self-efficacy score for each group (change).
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Market | Control - Planning
Number analyzed (Participants) | 251 | 166
score on a scale | 0.84 (1.04) | 1.37 (1.28)
Statistical Analysis 1: Comparison: Intervention - Market vs Control - Planning; Test type: Other — We used generalized linear mixed model (GLMM) with random intercept to control for clustering within sites; p = 0.75, GLMM — The p-value applies to the mean difference in mean self-efficacy change scores between the intervention and control groups; Mean Difference (Net) = -0.53, Standard Error of Mean 1.65

5. Other Pre Specified Outcome: Psychosocial Measures - Benefits (Expectations)
Description: Benefits (expectations) and barriers to eating F&V were measured with 12 questions using a 4-point Likert scale (1 indicates strongly disagree, 2 indicates disagree, 3 indicates agree, and 4 indicates strongly agree) previously tested in lower-income adults which reflects common benefits/barriers found in the literature. The 12 individual question scores were summed to generate the total barriers score, with a minimum score of 12 (strongly disagree) and a maximum score of 48 (strongly agree). For all scales, a higher number indicates higher perceived barriers and therefore a worse outcome. The lower the score the better the outcome.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention - Market | Control - Planning
Number analyzed (Participants) | 92 | 53
score on a scale | -0.32 (0.73) | 0.23 (0.86)
Statistical Analysis 1: Comparison: Intervention - Market vs Control - Planning; Test type: Other — We used generalized linear mixed model (GLMM) with random intercept to control for clustering within sites; p = 0.63, GLMM — P-value applies to the mean difference in mean total barriers score change between the intervention and control groups; Mean Difference (Net) = -0.56, Standard Error of Mean 1.13

ADVERSE EVENTS:
Time Frame: 1 year
Description: This is a low risk study. We do not anticipate any harm to the participants. Study staff reported adverse events to the PI within 24 hours and the PI reported all adverse events in accordance with the policy of the UB IRB. Because of this low risk status, the data safety monitoring plan (DSMP) focused on close monitoring, along with prompt reporting of excessive adverse events and any serious adverse events to the NIH and to the IRB. Recruitment, drop-out, and missing data will be reviewed.
Arm/Group | Intervention - Market | Control - Planning
All-Cause Mortality (participants affected / at risk) | 0/426 | 0/273
Serious Adverse Events (participants affected / at risk) | 0/426 | 0/273
Other Adverse Events (participants affected / at risk) | 0/426 | 0/273

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT04246593/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT04246593/SAP_001.pdf